CLINICAL TRIAL: NCT01670279
Title: A Phase 1, Multicenter, Randomized, Double-blind, Sequential Cohort, Placebo-controlled Trial to Assess the Safety and Tolerability of Ascending Multiple Oral Doses of Brexpiprazole as Adjunctive Therapy in the Treatment of Elderly Subjects With Major Depressive Disorder
Brief Title: Phase 1 Study to Assess the Safety/Tolerability of Brexpiprazole as Adjunctive Therapy in Elderly Subjects With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 331-12-291
Record Dates: First submitted 2012-08-07; First posted 2012-08-22 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 14 day titration phase and two fixed dose phases. The first fixed dose phase is 14 days with a daily dose of 2mg brexpiprazole/placebo. The second fixed dose phase is 14 days with a daily dose of 3 mg brexpiprazole/placebo.
  Interventions: Drug: Brexpiprazole
- Cohort 2 (Experimental): 14 day titration phase and a 14 day fixed dose phase a daily dose of 3mg brexpiprazole/placebo.
  Interventions: Drug: Brexpiprazole
- Cohort 3 (Experimental): 21 day titration phase and a 14 day fixed dose phase a daily dose of 3mg brexpiprazole/placebo.
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — up to 3mg oral dose once daily
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ascending multiple oral doses of brexpiprazole as adjunctive therapy in the treatment of elderly subjects with MDD.

DETAILED DESCRIPTION:
This is a phase 1, multicenter, randomized, double-blind, placebo-controlled, multiple ascending dose trial in 3 sequential cohorts of elderly subjects (age 70 to 85 years old) with MDD. Brexpiprazole will be administered as an adjunct treatment to the current antidepressant therapy that the subject is receiving. Total individual subject duration is expected to be no more than 119 days (a 30-day screening period, a 14-day washout period, up to 45-day in-clinic treatment period, and a 30-day follow-up after the last dose of trial medication).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent
* Ability to understand the nature of the trial and follow protocol requirements
* Male and female patients 70 to 85 years of age
* Subjects with normal or clinically stable findings on physical examination, medical history, clinical laboratory determinations, ECGs in relation to age
* BMI of 18 to 35 kg/m2.
* Stable subjects with a principal psychiatric diagnosis of MDD
* Subjects willing to discontinue all prohibited psychotropic and other prohibited medication

Exclusion Criteria:

* Sexually active males who are not practicing 2 different methods of birth control during the trial and for 30 days after the last dose of trial medication or who will not remain abstinent during the trial and for 30 days after the last dose
* Subjects who have had a vagus nerve stimulation device implanted or who have received ECT within 6 months of Screening
* Subjects with a current Axis I (DSM-IV-TR) diagnosis of:

  * Delirium, dementia, amnestic, or other cognitive disorder
  * Eating disorder (including anorexia nervosa or bulimia)
  * Obsessive-compulsive disorder
  * Panic disorder
  * Posttraumatic stress disorder or current or prior Axis I (DSM-IV-TR) diagnosis of Schizophrenia, schizoaffective disorder, or other psychotic disorder, Bipolar I or II disorder or bipolar disorder not otherwise specified
* Subjects with a clinically significant current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder
* Subjects experiencing hallucinations, delusions, or any psychotic symptomatology
* Subjects who have Active Suicidal Ideation with Some Intent to Act and whose most recent episode occurred within the last 6 months
* Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days
* Subjects with hypothyroidism or hyperthyroidism and/or an abnormal result for free T4 at Screening
* Subjects who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders
* Subjects with IDDM
* Subjects with uncontrolled hypertension (DBP > 95 mmHg) or symptomatic hypotension
* Subjects with epilepsy, a history of epilepsy, or a history of seizure
* Subjects with a positive drug screen for cocaine or other drugs of abuse
* The following laboratory test and ECG results are exclusionary:

  1. Platelets ≤ 75,000/mm3
  2. Hemoglobin ≤ 9 g/dL
  3. Neutrophils, absolute ≤ 1000/mm3
  4. AST > 3 × upper limit of normal
  5. ALT > 3 × upper limit of normal
  6. Creatinine ≥ 2 mg/dL
  7. HbA1c ≥ 7%
  8. QTcF ≥ 450 msec
* Treatment with a MAOI within the 2 weeks prior to the first dose of trial medication
* Use of benzodiazepines and/or hypnotics within 1 week prior the first dose of trial medication
* Use of oral neuroleptics within 30 days prior to or long-acting approved neuroleptics ≤ 1 full cycle plus 14 days prior to the first dose of trial medication on Day 1
* Prohibited concomitant medications used prior to randomization or anticipated need for such medications during the trial
* Subjects who would be likely to require prohibited concomitant therapy during the trial
* Subjects who received brexpiprazole in any prior clinical trial
* Subjects with a history of neuroleptic malignant syndrome
* Subjects with a history of true allergic response to more than 1 class of medications
* Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
* Subjects who participated in a clinical trial within the last 180 days or who participated in more than 2 clinical trials within the past year.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M. Youakim, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (4):
- United States (4):
  - Accurate Clinical Trials, Kissimmee, Florida
  - Miami Jewish Health System, Miami, Florida
  - St. Louis Clinical Trials, St Louis, Missouri
  - CRI Lifetree- Philadelphia Research Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 1, multicenter, randomized, double-blind, placebo-controlled, multiple ascending dose trial planned in 3 sequential cohorts of elderly participants (70 to 85 years old) with major depressive disorder (MDD). Brexpiprazole was administered as an adjunct treatment to the current antidepressant therapy that the participant received.
Pre-assignment Details: The study included a 30-day screening period, a 14-day washout period, up to 45-day inpatient treatment period (titration: received brexpiprazole or placebo once daily [QD] for 14 or 21 days and fixed dose phase: received assigned fixed dose for 14 or 28 days), and a 30-day follow-up after the last dose of study drug.
Groups:
- Brexpiprazole-Cohort 1: In the titration phase, participants received 0.5 mg brexpiprazole QD for 7 days, followed by 1 mg brexpiprazole QD for 7 days. In the fixed dose phase, participants received 2 mg brexpiprazole QD for 14 days, followed by 3 mg brexpiprazole QD for 14 days.
- Brexpiprazole-Cohort 2: In the titration phase, participants received 0.5 mg brexpiprazole QD for 7 days, followed by 1 mg brexpiprazole QD for 7 days. In the fixed dose phase, participants received 3 mg brexpiprazole QD for 14 days.
- Brexpiprazole-Cohort 3: In the titration phase, participants were to receive 0.5 mg brexpiprazole or placebo QD for 7 days, followed by 1 mg brexpiprazole or placebo QD for 7 days, and then 2 mg brexpiprazole or placebo QD for 7 days. In the fixed dose phase, participants were to receive 3 mg brexpiprazole or placebo QD for 14 days. However, Cohort 3 was not conducted due to safety and tolerability results from Cohorts 1 and 2.
- Placebo: In the titration phase, participants received 0.5 mg placebo QD for 7 days, followed by 1 mg placebo QD for 7 days. In the fixed dose phase, Cohort 1: participants received 2 mg placebo QD for 14 days, followed by 3 mg placebo QD for 14 days. Cohort 2: participants received 3 mg placebo QD for 14 days.
Period: Overall Study
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Brexpiprazole-Cohort 3 | Placebo
Started | 6 | 7 | 0 | 5
Completed | 6 | 5 | 0 | 4
Not Completed | 0 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Participant met withdrawal criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (4.0) | 76.0 (5.3) | 72.6 (1.5) | 74.1 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 13
  Male | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Tolerated Brexpiprazole
Description: Safety and tolerability of brexpiprazole was noted to be primary outcome measure. Brexpiprazole was judged to be tolerated if at least 6 out of 8 (75%) of the participants in a test cohort tolerated the dose after 14 days of QD dosing at the end of the fixed dose phase based on the blinded data. Dose toleration was defined as follows: during the course of the trial, the participants did not experience any moderate or severe adverse events (AEs) or potentially clinically relevant changes from Baseline in laboratory values, vital signs, electrocardiogram (ECG) tracings, Columbia-Suicide Severity Rating Scale (C-SSRS), or extrapyramidal symptom (EPS) ratings, which were assessed as possibly related to the study drug, and would have warranted a dose decrease or discontinuation of the study drug. The safety and tolerability of brexpiprazole was defined by parameters: AEs, laboratory values, vital signs, ECG, C-SSRS, or EPS ratings, the results of each of the parameters reported separately.
Time Frame: 45 Days
Population: Tolerability assessed in phase 1 trial in healthy participants (18-45 years) with MDD as adjunct therapy to ADTs; the efficacy assessed in phase 3 trials in participants (18-65 years) with MDD as adjunct therapy to ADTs. Thus, safety/tolerability of brexpiprazole in participants (>65 years) with MDD as adjunct therapy to ADTs was not characterized.
Measure: Number; unit: participants
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 7 | 5
participants | 6 | 7 | 5

2. Primary Outcome: Number of AEs Reported.
Description: The AEs were one of the primary parameters to measure the safety and tolerability of individual participants. The AEs were captured for all participants from the time the ICF was signed until the end of the trial. AEs were measured throughout the 14-day titration and 28-day fixed dose phase until follow-up (30 [±2] days after last dose of study medication).
Time Frame: Throughout the study, up to 119 days
Population: The safety dataset included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Events
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Events
  Adverse events | 12 | 33 | 5
  Treatment emergent adverse events (TEAEs) | 6 | 6 | 3
  Serious adverse events | 0 | 0 | 0

3. Primary Outcome: Incidence of Laboratory Values of Potential Clinical Significance
Description: The laboratory values were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria.
Time Frame: Titration Day 7, Fixed dose Day 14 and 28 and Last Visit
Population: The safety dataset included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Participants
  Cholesterol, fasting | 0 | 1 | 1
  Glucose | 0 | 0 | 1
  LDL direct, fasting | 0 | 0 | 1
  Triglycerides, fasting | 2 | 1 | 3
  Uric acid | 0 | 0 | 1
  Hematocrit | 0 | 2 | 1
  Prolactin | 2 | 0 | 0

4. Primary Outcome: Incidence of Vital Signs of Potential Clinical Significance
Description: The vital signs were one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance included abnormal values in heart rate, systolic and diastolic blood pressure, respiratory rate and weight that were identified based on pre-defined criteria.
Time Frame: Baseline, Titration Day 1, 2, 7, 8, Fixed Days 1, 2, 14, 15, 28, 29, Early Termination and Last Visit.
Population: The safety dataset included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Participants
  Weight increase | 2 | 0 | 0
  Supine hypotension, decrease | 1 | 0 | 0

5. Primary Outcome: Incidence of ECG Evaluations of Potential Clinical Significance
Description: The measurement of ECG was one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in heart rate and ECG intervals of PR, QRS, QT, QTcB, and QTcF that were identified based on pre-defined criteria.
Time Frame: Titratrion Day 1 and 7, Fixed dose Day 1, 14, 28, Early Termination
Population: The safety dataset included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Participants
  Supraventricular premature beat | 0 | 2 | 1
  Ventricular premature beat | 3 | 0 | 1
  Left bundle-branch block | 0 | 0 | 1
  Myocardial ischemia | 1 | 0 | 0
  Symmetrical T-wave inversions | 1 | 1 | 0
  Increase in QTcB | 1 | 3 | 2
  Increase in QTcF | 1 | 2 | 2

6. Primary Outcome: Incidence of Physical Examination Evaluation of Potential Clinical Significance
Description: The physical examination evaluation was one of the primary parameters to measure the safety and tolerability of individual participants. Incidence of TEAEs of potential clinical relevance include abnormal changes in the following body systems: head, ears, eyes, nose, and throat; thorax; abdomen; urogenital; extremities; neurological; and skin and mucosae.
Time Frame: Physical examination was performed at Screening, check-in, and discharge
Population: Safety Sample was analyzed. Any clinically significant condition present at the post-treatment physical examination that was not present at the baseline examination was documented as an adverse event and followed to a satisfactory conclusion. There were no clinically significant physical examination findings reported in this study.
Measure: Number; unit: Participants
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 0 | 0

7. Primary Outcome: Mean Change From Baseline to Study Completion in Simpson-Angus Scale (SAS) Total Score
Description: EPS was one of the primary parameters to measure the safety and tolerability of individual participants. The SAS is a rating scale used to measure EPS. The SAS scale consists of a list of 10 symptoms of parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia), with each item rated from 0 to 4, with 0 being normal and 4 being the worst. The SAS Total score is sum of ratings for all 10 items, with possible Total scores from 0 to 40.
Time Frame: End of Titration, Day 15, Day 29, Early Termination and Last visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Units on a scale
  End of Titration (N= 6, 6, 4) | -0.3 (0.5) | -0.5 (0.8) | -1.0 (0.8)
  Day 15 (N= 0, 5, 2) | NA (NA) — N=0, data not collected. | 0.2 (0.4) | -1.5 (0.7)
  Day 29 (N=6, 0, 2) | -0.3 (0.4) | NA (NA) — N=0, data not collected. | 0.0 (0.0)
  Early Termination (N= 0, 1, 1) | NA (NA) — N=0, data not collected. | -1.0 (NA) — N=1, standard deviation is not applicable. | 0.0 (NA) — N=1, standard deviation is not applicable.
  Last visit (N= 6, 6, 5) | -0.2 (0.4) | 0.0 (0.6) | -0.6 (0.9)

8. Primary Outcome: Mean Change From Baseline to Study Completion in Barnes Akathisia Global Score
Description: EPS was one of the primary parameters to measure the safety and tolerability of individual participants. The Barnes Akathisia Rating Scale was an EPS rating scale. The Barnes Akathisia Rating Scale was used to assess the presence and severity of akathisia. This scale consists of 4 items. Only the 4th item, the Global Clinical Assessment of Akathisia, was evaluated in this trial. This item is rated on a 6 point scale, with 0 being best (absent) and 5 being worst (severe akathisia).
Time Frame: End of Titration, Day 15, Day 29, Early Termination and Last visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Units on a scale
  End of Titration (N= 6, 6, 4) | -0.2 (0.4) | 0.0 (0.0) | -0.5 (0.6)
  Day 15 (N= 0, 5, 2) | NA (NA) — N=0, data not collected. | 0.0 (0.0) | -0.5 (0.7)
  Day 29 (N= 6, 0, 2) | 0.0 (0.0) | NA (NA) — N=0, data not collected. | -0.5 (0.7)
  Early Termination (N= 0, 1, 1) | NA (NA) — N=0, data not collected. | 0.0 (NA) — N=1, standard deviation is not applicable. | 0.0 (NA) — N=1, standard deviation is not applicable.
  Last visit (N= 6, 6, 5) | 0.0 (0.0) | 0.0 (0.0) | -0.4 (0.5)

9. Primary Outcome: Mean Change From Baseline to Study Completion in Abnormal Involuntary Movement Scale (AIMS) Rating Score.
Description: EPS was one of the primary parameters to measure the safety and tolerability of individual participants. The AIMS Scale was an EPS rating scale. The AIMS is a 12 item scale. The first 10 items are rated from 0 to 4 (0=best, 4=worst). Items 11 and 12, related to dental status, have dichotomous responses, 0=no and 1=yes. The AIMS Total Score is the sum of the ratings for the first seven items. The possible total scores are from 0 to 28.
Time Frame: End of Titration, Day 15, Day 29, Early Termination and Last visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Units on a scale
  End of Titration (N= 6, 6, 4) | 0.0 (0.0) | 0.2 (0.4) | 0.0 (0.0)
  Day 15 (N= 0, 5, 2) | NA (NA) — N=0, data not collected. | 0.0 (0.0) | 0.0 (0.0)
  Day 29 (N= 6, 0, 2) | 0.0 (0.0) | NA (NA) — N=0, data not collected. | 0.0 (0.0)
  Early Termination (N= 0, 1, 1) | NA (NA) — N=0, data not collected. | 0.0 (NA) — N=1, standard deviation is not applicable. | 0.0 (NA) — N=1, standard deviation is not applicable.
  Last Visit (N= 6, 6, 5) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

10. Primary Outcome: Change From Baseline to Study Completion in C-SSRS Score.
Description: The C-SSRS was one of the primary parameters to measure the safety and tolerability of individual participants. Suicidality was monitored during the trial using the C-SSRS. This scale consists of a baseline evaluation that assesses the lifetime experience of the participant with suicide events and suicidal ideation and a post-baseline evaluation that focuses on suicidality since the last trial visit.
Time Frame: Baseline, End of Titration, Fixed dose Day 14 and 28, Day 15 and 29, Early Termination, Last Visit
Population: Safety Sample includes all randomized participants who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Number analyzed (Participants) | 6 | 6 | 5
Participants
  Suicidality | 0 | 0 | 0
  Suicidal behaviour | 0 | 0 | 0
  Suicidal ideation | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were captured for all participants from the signing of the informed consent and were measured throughout the 14-day titration period, 28-day fixed dose period until follow-up (30 [±2] days after last dose of study medication).
Description: Participants who had received at least one dose of study medication were included in safety analysis.
Arm/Group | Brexpiprazole-Cohort 1 | Brexpiprazole-Cohort 2 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole-Cohort 1 (N=6) | Brexpiprazole-Cohort 2 (N=6) | Placebo (N=5)
Atrioventricular block first degree (Cardiac disorders) | 1 | 1 | 0
Hyperprolactinaemia (Endocrine disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Eye pruritis (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Blood pressure (Investigations) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Cohort 3 was not initiated based on the safety/tolerability results from Cohorts 1 and 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No